CLINICAL TRIAL: NCT06400979
Title: Aromatherapy for Management of Pain, Anxiety, and Nausea in the Acute Care Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Beekley Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1636824
Record Dates: First submitted 2024-01-06; First posted 2024-05-06 (Actual); Results first posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-03

CONDITIONS: Effectiveness of Aromatherapy
Keywords: aromatherapy; acute care unit; medical surgical unit; inhaled aromatherapy

STUDY DESIGN:
Intervention Model Description: To collect a sample of one hundred adult patients admitted to an acute care medical surgical unit. A quasi-experimental study with a single-arm pre-/post-test design evaluated one-time use of inhaled aromatherapy on hospitalized adults on an acute care unit. Pre-test tools included a numeric pain rating scale, facial anxiety scale and 0-5 nausea scale by Halpin et al. Aromatherapy (Elequil aromatabs) was administered for 8 hours. Sleep, satisfaction, well-being, and concurrent medication use were assessed post-aromatherapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Aromatherapy aromatab (Experimental): Interventional aromatherapy tab used to deliver inhaled aromatherapy to participants
  Interventions: Device: Elequil aromatab

INTERVENTIONS:
Device: Elequil aromatab — Aromatherapy impregnated tab utilized to dispense inhaled scent for the study

SUMMARY:
The purpose of this interventional study is to investigate the effects of aromatherapy on an acute care unit and whether it is effective in decreasing physical or emotional stressors that occur as a hospitalized patient. This study aimed to expand the limited literature on aromatherapy use in hospitalized adults and its effectiveness in decreasing pain, anxiety, and nausea. The hypothesis was that use of aromatherapy would decrease pain, anxiety and nausea in hospitalized adults and increase patient satisfaction. While there is anecdotal evidence of its efficacy, few studies exist evaluating its effectiveness within peer-reviewed journals, specifically on acute care medical surgical units.

DETAILED DESCRIPTION:
The goal for the study was to collect a sample of one hundred adult patients admitted to an acute care medical surgical unit. A quasi-experimental study with a single-arm pre-/post-test design evaluated one-time use of inhaled aromatherapy on hospitalized adults on an acute care unit. Pre-test tools included a numeric pain rating scale, facial anxiety scale and Halpin's 0-5 nausea scale. Aromatherapy (Elequil aromatabs) was administered for 8 hours. Sleep, satisfaction, well-being, and concurrent medication use were assessed post-aromatherapy. Descriptive and inferential statistics were performed. These subjects had to be conscious, oriented, able to consent, and able to understand the purpose of the study. Exclusion criteria were otolaryngology free flap patients (as this was a study being conducted on an otolaryngology acute care unit and another study was occurring with this population), patients with known allergies to essential oils, those taking sleep medications, or who have an aroma/essential oil contraindication. The use of a pre and post survey was used to measure the effectiveness of aromatherapy on pain, anxiety, and nausea. A baseline assessment was made of these ailments via Qualtrix. Subjects chose the aromatherapy tab fragrance that best fit their chief complaint, which was placed on their gown. After eight hours, a post-application survey to assess pain, anxiety, nausea, sleep/relaxation, overall satisfaction, and overall wellbeing was administered via Qualtrix. A numeric pain scale from 0-10, a 0-5 Likert Anxiety scale and a 0-5 nausea scale were used to measure efficacy. Sleep, satisfaction, and wellbeing was assessed with yes/no. A chart review to determine any measurable benefits in the reduction of related medications while using aromatherapy was to be conducted once one hundred subjects were obtained. The period for this study was approximately fifteen months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older,
* Admission to Tower 4 for an anticipated inpatient stay >24 hours,
* Alert and oriented,
* Capable of using a visual scale to self-report symptoms,
* Naïve to the use of aromatherapy for the use of decreasing pain, anxiety and/or nausea to participate,
* Not on a pediatric service.

Exclusion Criteria:

* Cognitively impaired,
* Post-op from an otolaryngologic surgery (another study was being conducted concurrently with this patient population and we did not want to interfere with those results),
* Known impaired olfactory function (limited or no sense of smell),
* On any psychiatric holds (e.g., 5150's),
* Known allergies to essential oils,
* Sensitive or allergic to plants (specifically to lavender plants, orange blossoms, sandalwood trees, or peppermint leaves) as essential oils are natural aromas derived from plants,
* Active participant of another Research Protocol,
* Admitted as a "short stay" or on "observation" status,
* Have a known history of Atrial Fibrillation. The use of peppermint has known effects on stimulating atrial fibrillation,
* Is a prisoner,
* Known pregnancy, or
* Expected to be transferred out of Tower 4 and/or discharged from the hospital within twenty-four hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UC Davis Medical Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No
We will not be sharing subject data after the conclusion of the study

REFERENCES:
- [Result] Frosch PJ, Johansen JD, Menne T, Pirker C, Rastogi SC, Andersen KE, Bruze M, Goossens A, Lepoittevin JP, White IR. Further important sensitizers in patients sensitive to fragrances. Contact Dermatitis. 2002 Nov;47(5):279-87. doi: 10.1034/j.1600-0536.2002.470204.x. PMID 12534532
- [Result] Bingham LJ, Tam MM, Palmer AM, Cahill JL, Nixon RL. Contact allergy and allergic contact dermatitis caused by lavender: A retrospective study from an Australian clinic. Contact Dermatitis. 2019 Jul;81(1):37-42. doi: 10.1111/cod.13247. Epub 2019 Apr 16. PMID 30779160
- [Result] Boehm K, Bussing A, Ostermann T. Aromatherapy as an adjuvant treatment in cancer care--a descriptive systematic review. Afr J Tradit Complement Altern Med. 2012 Jul 1;9(4):503-18. doi: 10.4314/ajtcam.v9i4.7. eCollection 2012. PMID 23983386
- [Result] Buckle J. The role of aromatherapy in nursing care. Nurs Clin North Am. 2001 Mar;36(1):57-72. PMID 11342402
- [Result] Johnson JR, Rivard RL, Griffin KH, Kolste AK, Joswiak D, Kinney ME, Dusek JA. The effectiveness of nurse-delivered aromatherapy in an acute care setting. Complement Ther Med. 2016 Apr;25:164-9. doi: 10.1016/j.ctim.2016.03.006. Epub 2016 Mar 7. PMID 27062964
- [Result] Cho MY, Min ES, Hur MH, Lee MS. Effects of aromatherapy on the anxiety, vital signs, and sleep quality of percutaneous coronary intervention patients in intensive care units. Evid Based Complement Alternat Med. 2013;2013:381381. doi: 10.1155/2013/381381. Epub 2013 Feb 17. PMID 23476690
- [Result] Cooke B, Ernst E. Aromatherapy: a systematic review. Br J Gen Pract. 2000 Jun;50(455):493-6. PMID 10962794
- [Result] Halpin A, Huckabay LM, Kozuki JL, Forsythe D. Weigh the benefits of using a 0-to-5 nausea scale. Nursing. 2010 Nov;40(11):18-20. doi: 10.1097/01.NURSE.0000389030.33760.7a. No abstract available. PMID 20975423
- [Result] Lakhan SE, Sheafer H, Tepper D. The Effectiveness of Aromatherapy in Reducing Pain: A Systematic Review and Meta-Analysis. Pain Res Treat. 2016;2016:8158693. doi: 10.1155/2016/8158693. Epub 2016 Dec 14. PMID 28070420
- [Result] Lis-Balchin M. Essential oils and 'aromatherapy': their modern role in healing. J R Soc Health. 1997 Oct;117(5):324-9. doi: 10.1177/146642409711700511. PMID 9519666
- [Result] Long L, Huntley A, Ernst E. Which complementary and alternative therapies benefit which conditions? A survey of the opinions of 223 professional organizations. Complement Ther Med. 2001 Sep;9(3):178-85. doi: 10.1054/ctim.2001.0453. PMID 11926432
- [Result] Maddocks-Jennings W, Wilkinson JM. Aromatherapy practice in nursing: literature review. J Adv Nurs. 2004 Oct;48(1):93-103. doi: 10.1111/j.1365-2648.2004.03172.x. PMID 15347415
- [Result] Moeini M, Khadibi M, Bekhradi R, Mahmoudian SA, Nazari F. Effect of aromatherapy on the quality of sleep in ischemic heart disease patients hospitalized in intensive care units of heart hospitals of the Isfahan University of Medical Sciences. Iran J Nurs Midwifery Res. 2010 Fall;15(4):234-9. PMID 22049287
- [Result] Quinlan-Colwell AD. Understanding the paradox of patient pain and patient satisfaction. J Holist Nurs. 2009 Sep;27(3):177-82; quiz 183-5. doi: 10.1177/0898010109332758. Epub 2009 Jul 8. PMID 19587387
- [Result] Shin BC, Lee MS. Effects of aromatherapy acupressure on hemiplegic shoulder pain and motor power in stroke patients: a pilot study. J Altern Complement Med. 2007 Mar;13(2):247-51. doi: 10.1089/acm.2006.6189. PMID 17388768
- [Result] Vickers A. Yes, but how do we know it's true? Knowledge claims in massage and aromatherapy. Complement Ther Nurs Midwifery. 1997 Jun;3(3):63-5. doi: 10.1016/s1353-6117(97)80035-2. PMID 9439251
- See also: Instructional video on how to use aromatab — https://vimeo.com/276457486

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study took place from December 1, 2020 to May 1, 2022.This study aimed to collect a sample of one hundred adult patients admitted to an acute care medical surgical unit.
Pre-assignment Details: Ninety-four subjects of the intended one hundred were enrolled and consented. Sixty-four completed the study in its entirety, with both pre- and post-surveys being administered. Reasons for not having a post-survey completed: lack of communication of when the post- survey should be given, patient was asleep, no investigator working to administer the post-test, or the post-test was simply forgotten. One participant did not complete the study because it was stated that the scent was too strong.
Groups:
- Aromatherapy Aromatab: Interventional aromatherapy tab used to deliver inhaled aromatherapy to participants
  The study used an Elequil aromatab which is an aromatherapy impregnated tab utilized to dispense a specific inhaled scent for the study. Each aromatherapy tab was used to determine its effects on pain, nausea and anxiety.
Period: Overall Study
Arm/Group | Aromatherapy Aromatab
Started | 94
Completed | 64
Not Completed | 30
Not completed — Lost to Follow-up | 29
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Of the 94 consented subjects, 64 subjects completed the study in its entirety, with both pre- and post-surveys administered.
Groups:
- Aromatherapy Aromatab: Interventional aromatherapy tab used to deliver inhaled aromatherapy to participants
  Use of an Elequil aromatab which is an aromatherapy impregnated tab utilized to dispense inhaled scent for the study. Each tab is impregnated with a specific essential oil that corresponds to either pain, anxiety or nausea.
Arm/Group | Aromatherapy Aromatab
Number analyzed (Participants) | 94
Age, Customized [Count of Participants; unit: Participants]
  Age of Participant: >18 to 65 | 80
  Age of Participant: >65 | 14
Sex/Gender, Customized [Number; unit: participants]
  Female | 59
  Male | 35
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Numerical Rating Pain Scale
Description: The Numerical Rating Pain Scale measures pain experienced right now based on a 11-point Likert scale with choices of 0 = no pain, 5 = Moderate pain, 10 = Worst possible pain.
Time Frame: Pre-Post Aromatherapy Administration (8 hours)
Population: Number of subjects utilizing aromatherapy tabs to decrease pain
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Aromatherapy Aromatab: Interventional aromatherapy tab used to deliver inhaled aromatherapy to participants
  Elequil aromatab: Aromatherapy impregnated tab utilized to dispense inhaled scent for the study to analyze the effectiveness in decreasing pain.
Arm/Group | Aromatherapy Aromatab
Number analyzed (Participants) | 94
score on a scale
  Pre-score for subjects utilizing Aromatherapy for pain | 5.7 (3.0)
  Post-score for subjects utilizing Aromatherapy for symptom management for pain: number analyzed (Participants) | 64
  Post-score for subjects utilizing Aromatherapy for symptom management for pain | 5.3 (2.9)
  Pain: Post vs Pre: number analyzed (Participants) | 64
  Pain: Post vs Pre | -1 (2.9)
Statistical Analysis 1: Comparison: Aromatherapy Aromatab; Test type: Superiority; p = 0.008, ANCOVA

2. Primary Outcome: Nausea Scale
Description: Nausea Scale: 0-5 Nausea Scale. 0 - No nausea and 5 - severe nausea
Time Frame: Pre-Post Aromatherapy Administration (8 hours)
Population: Total number of subjects participating in the study
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Aromatherapy Aromatab: Interventional aromatherapy tab used to deliver inhaled aromatherapy to participants
  Elequil aromatab: Aromatherapy impregnated tab utilized to dispense inhaled scent for the study to analyze the effectiveness in decreasing nausea
Arm/Group | Aromatherapy Aromatab
Number analyzed (Participants) | 94
score on a scale
  Pre-score for subjects utilizing aromatherapy to decrease nausea: number analyzed (Participants) | 93
  Pre-score for subjects utilizing aromatherapy to decrease nausea | 1.5 (1.7)
  Post-score for subjects utilizing aromatherapy for symptom management for nausea: number analyzed (Participants) | 56
  Post-score for subjects utilizing aromatherapy for symptom management for nausea | 1.2 (1.6)
Statistical Analysis 1: Comparison: Aromatherapy Aromatab; Test type: Superiority — To assess the reduction of nausea following aromatherapy, pre- and post- aromatherapy scores were compared using paired t-tests; p = 0.13, ANCOVA

3. Primary Outcome: Anxiety Likert Scale
Description: This one-item scale consisted of five evenly spaced numbers each anchored to a level of anxiety (0 = not at all anxious, 2 = a little anxious, 3 = moderately anxious, 4 = very anxious, 5 = extremely anxious).
Time Frame: Pre-Post Aromatherapy Admin (8 hours)
Population: Number of subjects utilizing aromatherapy to decrease anxiety.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aromatherapy Aromatab
Number analyzed (Participants) | 94
score on a scale
  Pre-score for subjects utilizing aromatherapy to decrease anxiety | 2.6 (1.9)
  Post-score for subjects utilizing aromatherapy for symptom management for anxiety: number analyzed (Participants) | 63
  Post-score for subjects utilizing aromatherapy for symptom management for anxiety | 1.8 (1.6)
Statistical Analysis 1: Comparison: Aromatherapy Aromatab; Test type: Superiority; p < 0.0001, ANCOVA

4. Secondary Outcome: Patient Satisfaction
Description: The use of a post-survey to evaluate effectiveness of aromatherapy on patient satisfaction using a yes or no response.
Time Frame: 8 hours
Population: Number of subjects utilizing aromatherapy to measure its effectiveness on patient satisfaction.
Measure: Count of Participants; unit: Participants
Groups:
- Aromatherapy Aromatab: Interventional aromatherapy tab used to deliver inhaled aromatherapy to participants
  The study used an Elequil aromatab which is an aromatherapy impregnated tab utilized to dispense a specific inhaled scent for the study. Each aromatherapy tab was used to determine its effects on pain, nausea and anxiety. In addition, subjects were asked to rate their level of satisfaction while being in the hospital.
Arm/Group | Aromatherapy Aromatab
Number analyzed (Participants) | 94
Participants
  Number of subjects utilizing aromatherapy resulting in an increase in patient satisfaction | 47
  Number of subjects utilizing aromatherapy resulting in a decrease in patient satisfaction | 17
  Number of unknown responses | 30
Statistical Analysis 1: Comparison: Aromatherapy Aromatab; Test type: Other — Perceived effectiveness of aromatherapy for patient satisfaction were compared with respect to post-aromatherapy scores and pre-post changes in scores using two-sample t-tests; p = 0.02, t-test, 2 sided

5. Secondary Outcome: Well-being
Description: The use of a post-survey to evaluate effectiveness of aromatherapy on the subject's well-being using a yes or no response.
Time Frame: 8 hours
Population: Number of subjects utilizing aromatherapy to measure its effectiveness on the subject's well-being.
Measure: Count of Participants; unit: Participants
Groups:
- Aromatherapy Aromatab: Interventional aromatherapy tab used to deliver inhaled aromatherapy to participants
  The study used an Elequil aromatab which is an aromatherapy impregnated tab utilized to dispense a specific inhaled scent for the study. Each aromatherapy tab was used to determine its effects on pain, nausea and anxiety. In addition
Arm/Group | Aromatherapy Aromatab
Number analyzed (Participants) | 94
Participants
  Number of subjects utilizing aromatherapy resulting in an increase in patient well-being | 50
  Number of subjects utilizing aromatherapy resulting in a decrease in patient well-being | 19
  Number of unknown responses | 25
Statistical Analysis 1: Comparison: Aromatherapy Aromatab; Test type: Superiority; p = 0.02, ANCOVA

6. Secondary Outcome: Increased Sleep
Description: The use of a post-survey to evaluate effectiveness of aromatherapy in increasing sleep using a yes or no response.
Time Frame: 8 hours
Population: Number of subjects utilizing aromatherapy to measure its effectiveness on sleep
Measure: Count of Participants; unit: Participants
Arm/Group | Aromatherapy Aromatab
Number analyzed (Participants) | 94
Participants
  Number of subjects utilizing aromatherapy to measure its effectiveness on increasing sleep. | 55
  Number of subjects utilizing aromatherapy resulting in a decrease in sleep. | 10
  Number of unknown responses. | 29
Statistical Analysis 1: Comparison: Aromatherapy Aromatab; Test type: Superiority; p = 0.02, ANCOVA

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for the duration of patient enrollment in the study (8 hours during hospitalization).
Groups:
- Aromatherapy Aromatab Used to Measure Effectiveness on Decreasing Pain: Interventional aromatherapy tab used to deliver inhaled aromatherapy to participants
  Elequil aromatab: Aromatherapy impregnated tab utilized to dispense inhaled scent for the study to analyze the effectiveness in decreasing pain. No adverse effects were noted
Arm/Group | Aromatherapy Aromatab Used to Measure Effectiveness on Decreasing Pain
All-Cause Mortality (participants affected / at risk) | 0/94
Serious Adverse Events (participants affected / at risk) | 0/94
Other Adverse Events (participants affected / at risk) | 0/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aromatherapy Aromatab Used to Measure Effectiveness on Decreasing Pain (N=94)
Dermatitis (General disorders) | 0 (0)
Runny nose/ nasal congestion (sinus issues) (General disorders) | 0 (0)
Rash (General disorders) | 0 (0)
Red or bumpy skin (indurations) (General disorders) | 0 (0)
Increased discomfort (General disorders) | 0 (0)
Anaphylactic symptoms (General disorders) | 0 (0)

LIMITATIONS AND CAVEATS:
Limitations included slow enrollment, study design and missing post-test scores. We had a slow start with enrolling subjects as many patients either did not fit the eligibility criteria, or they were not interested. In addition, with the COVID pandemic, it made it even more difficult to enroll patients. Finding our requisite number of subjects was more challenging than expected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-02-20): https://cdn.clinicaltrials.gov/large-docs/79/NCT06400979/Prot_002.pdf
  • Informed Consent Form (2020-09-18): https://cdn.clinicaltrials.gov/large-docs/79/NCT06400979/ICF_001.pdf